CLINICAL TRIAL: NCT00951600
Title: An Open Label, Balanced, Randomised, Two-treatment, Two-period, Two-sequence, Single-dose, Crossover Bioavailability Study Comparing Oxcarbazepine 300 mg/5mL Oral Suspension of OHM Laboratories (a Subsidiary of Ranbaxy Pharmaceuticals Inc) With Trileptal® 300 mg/5mL Oral Suspension (Containing Oxcarbazepine 300 mg/5mL) of Novartis Pharmaceutical Corporation in Healthy, Adult, Male, Human Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study of Oxcarbazepine Oral Suspension 300 mg/5 mL Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 228_OXCAR_06
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Oxcarbazepine oral suspension fasting study
MeSH Terms: interventions — Oxcarbazepine; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Oxcarbazepine oral suspension 300 mg/5mL of OHM Laboratories Inc. (a subsidiary of Ranbaxy Pharmaceuticals Inc.)
  Interventions: Drug: oxcarbazepine 300 mg/5mL oral suspension
- 2 (Active Comparator): Trileptal® (oxcarbazepine) oral suspension 300 mg/5mL of Novartis
  Interventions: Drug: oxcarbazepine 300 mg/5mL oral suspension

INTERVENTIONS:
Drug: oxcarbazepine 300 mg/5mL oral suspension

SUMMARY:
The study was conducted as an open label, balanced, randomized, two-treatment, two-period, two-sequence, single- dose, crossover bioavailability study comparing oxcarbazepine 300 mg/5mL oral suspension of OHM Laboratories (a subsidiary of Ranbaxy Pharmaceuticals Inc.) with Trileptal® 300 mg/5mL oral suspension (containing oxcarbazepine 300 mg/5mL) of Novartis Pharmaceutical Corporation in healthy, adult, male, human subjects under fasting conditions.

DETAILED DESCRIPTION:
Following an overnight fast of at least 10 hours, a single dose of 10 mL of oxcarbazepine 300 mg/5 mL oral suspension (containing oxcarbazepine 300 mg/5rnL) was administered using a 10 mL graduated syringe, during each period of the study under the supervision of trained study personnel, along with 240 mL of drinking water at ambient temperature.

During the course of the study safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical parameters, serology and urine analysis) at baseline. Laboratory parameters of hematology and biochemistry were repeated at the end of the study.

A total of forty (40) subjects were administered a single oral dose of the test or reference formulation of 10 mL of oxcarbazepine 300 mg/5 mL oral suspension (containing oxcarbazepine 300 mg/5mL) according to a randomization schedule. Thirty-five (35) subjects completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Were in the age range of 18-45 years.
2. Were neither overweight nor underweight for the corresponding height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
3. Had voluntarily given written informed consent to participate in this study
4. Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

There were no deviations in this regard.

Exclusion Criteria:

1. History of hypersensitivity to oxcarbazepine, carbamazepine or to any related drugs.
2. History of hyponatremia, diplopia.
3. Recent history of dizziness, somnolence, and abdominal pain.
4. Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
5. Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
6. Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for hemoglobin, total white blood cells count, differential WBC count or platelet count.
7. Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids).
8. Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
9. Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), glucose (positive) or protein (positive).
10. Clinically abnormal ECG or Chest X-ray.
11. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or hematological disease, diabetes or glaucoma.
12. History of any psychiatric illness, which might impair the ability to provide written informed consent.
13. Regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period.
14. History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or I glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
15. Use of any enzyme modifying drugs within 30 days prior to Day 1 of this study.
16. Participation in any clinical trial within 12 weeks preceding Day 1 of this study.
17. Subjects who, through completion of this study, had donated and/or lost more than 350 mL of blood in the past 3 months.

There were no deviations in this regard.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of ranbaxy Oxcarbazepine oral suspension 300 mg/5mL under fasting condition

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy Clinical Pharmacology Unit, Ranbaxy Laboratories Limited, Noida, Uttar Pradesh, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html